CLINICAL TRIAL: NCT02008942
Title: Reliable Inhibition of Thrombocyte Activity: Comparison of PL2200 Aspirin Capsules, 325 mg and Enteric-Coated Aspirin (RITE Study)
Brief Title: Pharmacodynamic Evaluation of PL2200 Versus Enteric-Coated Aspirin in Diabetic Patients
Acronym: RITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PL-ASA-006
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PL2200 Aspirin Capsules (Experimental): PL2200 Aspirin Capsules
  Interventions: Drug: PL2200 Aspirin Capsules
- Enteric-coated aspirin caplets (Active Comparator): Enteric-coated aspirin caplets
  Interventions: Drug: Enteric-coated aspirin caplets

INTERVENTIONS:
Drug: PL2200 Aspirin Capsules — 325 mg aspirin; once per day for 10 days
  Arms: PL2200 Aspirin Capsules
Drug: Enteric-coated aspirin caplets — 325 mg aspirin; once per day for 10 days
  Arms: Enteric-coated aspirin caplets

SUMMARY:
This study will determine if aspirin from PL2200, an investigational product, gets into the blood stream as quickly as enteric coated aspirin, and to test whether PL2200 is able to prevent blood clots as effectively as enteric coated aspirin, when administered to patients with diabetes

ELIGIBILITY:
Inclusion Criteria:

* Non-Insulin-Dependent Diabetes Mellitus
* Adults 21 to 79 years, inclusive
* Body mass index between 30 and 40 kg/m2, inclusive

Exclusion Criteria:

* Currently prescribed aspirin or anti-coagulants
* Contraindications to aspirin
* Significant disease history or active disease other than Non-Insulin-Dependent Diabetes Mellitus
* Patient requires insulin

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami Research Associates, Miami, Florida
  - PRA Clinical Pharmacology Center, Lenexa, Kansas
  - Medpace Clinical Pharmacology, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- PL2200 Aspirin First, Then Enteric Coated (EC) Aspirin: First Intervention Period:
  PL2200 Aspirin Capsules: 325 mg aspirin; once per day for 10 days
  (after 2-week washout period)
  Second Intervention Period:
  EC aspirin: 325 mg aspirin; once per day for 10 days
- Enteric Coated (EC) Aspirin First, Then PL2200 Aspirin: First Intervention Period:
  EC aspirin: 325 mg aspirin; once per day for 10 days
  (after 2-week washout period)
  Second Intervention Period:
  PL2200 Aspirin Capsules: 325 mg aspirin; once per day for 10 days
Period: First Intervention
Arm/Group | PL2200 Aspirin First, Then Enteric Coated (EC) Aspirin | Enteric Coated (EC) Aspirin First, Then PL2200 Aspirin
Started | 27 | 30
Completed | 27 | 30
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | PL2200 Aspirin First, Then Enteric Coated (EC) Aspirin | Enteric Coated (EC) Aspirin First, Then PL2200 Aspirin
Started | 26 | 30
Completed | 25 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients that received at least 1 dose of study drug
Groups:
- All Study Participants: All patients that received at least 1 dose of study drug
Arm/Group | All Study Participants
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Time to 99% Inhibition of Serum Thromboxane
Description: Serial measurements of aspirin anti-platelet activity will be collected over 11 days, and compared between groups, to allow a determination of pharmacodynamic (anti-platelet) bioequivalence between study drugs. Aspirin's antiplatelet activity is measured by the capacity of platelets to generate serum thromboxane (a surrogate marker for inhibition of COX-1 by aspirin). Inhibition of serum thromboxane is a key marker of antiplatelet efficacy.
Time Frame: 11 days
Population: Pharmacodynamic (PD) Evaluable Population - patients in the intent-to-treat population who received a full treatment regimen for each of 2 study drugs, had all scheduled PD blood draws, and had no other major protocol violations.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PL2200 Aspirin Capsules | Enteric-coated Aspirin Caplets
Number analyzed (Participants) | 55 | 55
hours | 26.71 (62.758) | 64.57 (72.842)

ADVERSE EVENTS:
Description: Intent-to-Treat Population: patients that received at least 1 dose of study drug.
Arm/Group | PL2200 Aspirin Capsules | Enteric-coated Aspirin Caplets
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 2/57 | 2/56
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PL2200 Aspirin Capsules (N=57) | Enteric-coated Aspirin Caplets (N=56)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard confidentiality agreement